CLINICAL TRIAL: NCT03198650
Title: A Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics and Anti-tumour Activity of Acalabrutinib, a Selective and Irreversible Bruton's Tyrosine Kinase Inhibitor, in Japanese Adult Patients With Advanced B-cell Malignancies
Brief Title: A Phase 1 Study of Acalabrutinib in Japanese Adult Patients With Advanced B-cell Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8220C00001
Record Dates: First submitted 2017-06-14; First posted 2017-06-26 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Part1: Advanced B-cell Malignancies; Part2: r/rCLL and r/rMCL; Part3: Untreated CLL
MeSH Terms: interventions — acalabrutinib; obinutuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1 / Part 2 (Experimental): Acalabrutinib
  Interventions: Drug: Acalabrutinib
- Part 3 (Experimental): Acalabrutinib in combination with Obinutuzumab
  Interventions: Drug: Acalabrutinib; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Acalabrutinib — Acalabrutinib
Drug: Obinutuzumab — Obinutuzumab
  Arms: Part 3

SUMMARY:
This is a multicenter, open-label Phase 1 study of acalabrutinib, a selective and irreversible Bruton's tyrosine kinase inhibitor, in Japanese adult patients with advanced B-cell malignancies. This study is divided into 3 parts: Part 1 (dose-confirmation phase), Part 2 (dose-expansion phase) and Part 3 (dose-confirmation phase for combination therapy).

ELIGIBILITY:
Key Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures, sampling and analyses
* Japanese subjects at least 20 years of age at the time of study entry.
* Presence of radiographically measurable lymphadenopathy or extranodal lymphoid malignancy (defined as the presence of a ≥ 2.0 cm lesion as measured in the longest dimension by computerised tomography [CT] scan). Note: Not applicable to subjects with Chronic lymphocytic leukemia (CLL), Waldenström macroglobulinemia (WM)
* Eastern Co-operative Oncology Group (ECOG) Performance Status (PS) of ≤ 2
* Adequate organ function defined as follows: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2 × institutional upper limit of normal (ULN), total bilirubin ≤ 1.5 × ULN except in the case of subjects with documented Gilbert's disease, ≤ 2.5 × ULN
* Serum amylase ≤1.5 × ULN or serum lipase ≤1.5 × ULN <Part2>
* Relapsed or refractory CLL/SLL: Confirmed diagnosis of CLL/SLL, which has relapsed after, or been refractory to ≥ 1 prior therapy for CLL/SLL, and has active disease meeting IWCLL 2008 criteria (Hallek 2008).
* Relapse or refractory MCL: Confirmed diagnosis of MCL, which has relapsed after,or been refractory to ≥ 1 prior therapy for MCL, and documented failure to achieve at least PR with, or documented disease progression after, the most recent treatment regimen.

<Part3>

* Japanese subjects:

  1. ≥ 65 years of age OR
  2. ≥ 20 and < 65 years of age, provided that they meet at least one of the following criteria:

  i. Creatinine clearance 30 to 69 mL/min using the Cockcroft-Gault equation. ii. A score higher that 6 on the Cumulative Illness Rating Scale-Geriatric
* Diagnosis of CD20+ CLL that meets published diagnostic criteria (Hallek 2008):

  1. Monoclonal B cells (either kappa or lambda light chain restricted) that are clonally co-expressing ≥ 1 B-cell marker (CD19, CD20, or CD23) and CD5.
  2. Prolymphocytes may comprise ≤ 55% of blood lymphocytes.
  3. Presence of ≥ 5000 μL B lymphocytes in the peripheral blood (at any point since diagnosis)

Key Exclusion Criteria:

* History of other invasive malignancy within 2 years except for cervical carcinoma in situ (CIS), non-melanomatous carcinoma of the skin or ductal carcinoma in situ (DCIS) of the breast that have been surgically cured.
* A life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of acalabrutinib, or put the study outcomes at undue risk
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification (New York Heart Association Functional Classification 1994).
* Malabsorption syndrome, disease significantly affecting GI function, resection of the stomach, extensive small bowel resection that is likely to affect absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery such as gastric bypass.
* Known CNS involvement by lymphoma/leukemia
* Known prolymphocytic leukemia or history of, or currently suspected, Richter's syndrome (for CLL/SLL)
* Receipt of any biological or immunological based therapies (including experimental therapies) for leukaemia or lymphoma or myeloma (including, but not limited to, MAb therapy such as rituximab, or cancer vaccine therapies) within 4 weeks prior to the first dose of acalabrutinib.
* Any prior therapy with BCR inhibitors (eg, BTK, PI3Kδ, or SYK inhibitors) or BCL-2 inhibitors (eg, venetoclax/ABT-199)
* Known history of HIV, serologic status reflecting active hepatitis B or C infection,or any uncontrolled active systemic infection.
* History of stroke or intracranial haemorrhage within 6 months prior to first dose of study drug.
* Ongoing, drug-induced liver injury, alcoholic liver disease, nonalcoholic steatohepatitis, primary biliary cirrhosis, ongoing extrahepatic obstruction caused by cholelithiasis, cirrhosis of the liver, or portal hypertension.
* History of or ongoing drug-induced pneumonitis
* Estimated creatinine clearance of < 30 mL/min, calculated using the formula of Cockcroft and Gault [(140-Age) • Mass (kg)/(72 • creatinine mg/dL); multiply by 0.85 if female]
* Significant screening electrocardiogram (ECG) abnormalities including left bundle-branch block, 2nd degree AV block type II, 3rd-degree AV block, Grade ≥ 2 bradycardia, and the average QT interval corrected for heart rate (QTc) from the three screening ECGs must be > 480 msec (calculated using Fridericia's formula: QT/RR0.33)
* Concurrent participation in another therapeutic clinical trial.
* History of bleeding diathesis (eg, hemophilia or von Willebrand disease)
* Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists (eg, phenprocoumon) within 7 days before first dose of study drug.
* Requires treatment with proton pump inhibitors (eg, omeprazole, esomeprazole, lansoprazole or rabeprazole). Subjects receiving proton pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrollment to this study.
* Presence of a GI ulcer diagnosed by endoscopy within 3 months before screening.
* Uncontrolled autoimmune hemolytic anemia (AIHA) or immune thrombocytopenic purpura (ITP).

Ages: 20 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs), Serious Adverse Events (SAEs) and dose-limiting toxicities (DLTs) as a measure of safety and tolerability. | From the first dose of study treatment to data cut-off date defined as 2 years after last subject enrolled. In Part 1, DLT will be evaluated in Cycle 1 (28 days). In Part 3, DLT will be evaluated in Cycle 2 (28 days).
  Acalabrutinib is considered as safe and tolerable if ≦1 of 6 patients experiences a DLT.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | From the date of first dose to Cycle 3 Day 28.
  Pharmacokinetics (PK) parameters will be derived using standard non-compartmental methods.
Free Bruton's Tyrosine Kinase (BTK) not occupied by acalabrutinib | From the date of first dose to end of treatment visit, up to 80 months
  Free BTK not occupied by acalabrutinib is measured and BTK occupancy at each timepoint is calculated relative to the predose timepoint. The signal of the predose sample represents 100% free BTK (0% occupied BTK), while each sample incubated with 1 μM exogenous acalabrutinib represents 0% free BTK (100% occupied BTK).
Overall response rate | From the start of acalabrutinib therapy to earlier of the first documentation of objective disease progression or death from any cause, whichever came first up to 80 months
  Defined as the proportion of subjects who achieve a response.
Duration of Response | From the start of acalabrutinib therapy to earlier of the first documentation of objective disease progression or death from any cause, whichever came first up to 80 months
  Defined as the interval from the first documentation of response to the earlier of the first documentation of definitive disease progression or death from any cause.
Progression free survival | From the start of acalabrutinib therapy to earlier of the first documentation of objective disease progression or death from any cause, whichever came first up to 80 months
  Defined as the interval from the start of acalabrutinib therapy to the earlier of the first documentation of objective disease progression or death from any cause.
Area under the plasma concentration-time curve (AUC) | From the date of first dose to Cycle 3 Day 28
  PK parameters will be derived using standard non-compartmental methods.
Time to Cmax (tmax) | From the date of first dose to Cycle 3 Day 28
  PK parameters will be derived using standard non-compartmental methods.

CONTACTS AND LOCATIONS:
Locations (13):
- Japan (13):
  - Research Site, Chiba
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Isehara-shi
  - Research Site, Izumo-shi
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Okayama
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shimotsuke-shi
  - Research Site, Suita-shi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Astra Zeneca Clinical Trials website — https://www.astrazenecaclinicaltrials.com/study/D8220C00001/